CLINICAL TRIAL: NCT05597345
Title: Selinexor for the Treatment of Patients with Intermediate and High-Risk Smoldering Multiple Myeloma
Brief Title: Selinexor for the Treatment of Intermediate and High-Risk Smoldering Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Brea Lipe, Professor - Department of Medicine , Hematology/Oncology (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMMMY22027
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Smoldering Multiple Myeloma; Smoldering Myeloma; Multiple Myeloma; Myeloma; MGUS
MeSH Terms: conditions — Smoldering Multiple Myeloma; Multiple Myeloma; Neoplasms, Plasma Cell | interventions — selinexor

STUDY DESIGN:
Intervention Model Description: This is a single-center, open-label, phase 2, single-arm clinical trial of selinexor in patients with intermediate to high-risk smoldering multiple myeloma. Intermediate-risk patients will start enrolling after 5 high-risk smoldering myeloma patients have been enrolled and received 1-2 cycles of treatment. Patients will receive selinexor 40mg orally weekly for up to 12 cycles. Each cycle will be 28 days in length. Patients will receive treatment up to 1 year and continue in follow-up for 2 years after completion of the treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Treatment (Experimental): Selinexor 40mg weekly for up to 12 cycles. Each cycle will be 28 days in length.
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — Low-dose Selinexor for the Treatment of Intermediate to High-Risk Smoldering Multiple Myeloma

SUMMARY:
Selinexor is a drug that has been approved in the treatment of patients with symptomatic multiple myeloma. The standard of care for patients with Smoldering Multiple Myeloma remains observation, but there are numerous clinical trials investigating interventions to delay progression to multiple myeloma and prevent or delay disease related outcomes. A subset of patients with intermediate or high risk smoldering multiple myeloma have a much higher risk of progressive to multiple myeloma, while the low risk smoldering myeloma patient population has a much lower risk. This is a clinical trial investigating the use of low-dose selinexor in patients with intermediate to high-risk smoldering multiple myeloma. The investigators hypothesize that the use of selinexor in intermediate to high risk smoldering myeloma patients will help to delay progression of disease to symptomatic multiple myeloma.

DETAILED DESCRIPTION:
Plasma cell disorders are a spectrum of diseases ranging from monoclonal gammopathy of undetermined significance (MGUS), to smoldering multiple myeloma (SMM), to multiple myeloma (MM). Multiple myeloma is preceded by an asymptomatic precursor state in the majority of cases. While the vast majority of these patients do not progress to have symptomatic disease, there is an intermediate to high-risk subset of patients with SMM that do go on to meet criteria for MM, including hypercalcemia, anemia, renal insufficiency, and lytic bone lesions.

There are numerous risk stratification systems that have been devised to predict which patients have the highest risk of progression. The Mayo Clinic group identified 3 factors as predictors for early progression. these factors include a bone marrow plasma cell burden of greater than 20%, a monoclonal protein (M-spike) of 2g/dL or greater, and a ratio of involved to uninvolved serum free light chains of 20% or greater. Patients with one more of these risk factors have an increased risk of progression to MM in the first five years after diagnosis.

The current standard of care for the treatment of patients with SMM is observation because numerous early studies failed to demonstrate a survival advantage with pharmacologic intervention. More recent studies have aimed to select out the high-risk patients where intervention is more likely to be beneficial in preventing or delaying progression. The approaches have ranged in intensity and aim, with some approaches aimed at preventing or delaying progression, and others aimed at treating aggressively with curative intent. While the preliminary results of these studies have been promising, there is no consensus on the optimal approach in patients with intermediate to high-risk smoldering multiple myeloma.

Selinexor is a small-molecule selective inhibitor of nuclear export (SINE), which inhibits exportin-1 (XPO1) in a slowly reversible, covalent manner. XPO1 is a transport protein that is responsible for transport of over 200 proteins from the nucleus to the cytoplasm. Inhibition of XPO1 leads to accumulation of tumor suppressor proteins, cell-cycle regulators, and oncoprotein mRNAs in the nucleus and eventually leads to apoptosis of malignant cells. XPO1 inhibition has been shown to induce apoptosis in malignant MM cells and impede osteoclastogenesis without toxicity to surrounding bone marrow stromal cells (BMSCs).

Selinexor has been FDA approved for the treatment of relapsed and refractory multiple myeloma and is currently being studied in the frontline and relapsed settings with different therapeutic combinations in the STOMP trial. Selinexor has not been studied in the precursor disease population. While the exact mechanisms of progression from SMM to MM are incompletely understood, it has been shown that XPO1 expression is increased during progression of disease, which makes this a promising target in this population of patients. The investigators aim to limit the side effect profile while maintaining efficacy of treatment for SMM, with the goal of delaying or preventing progression to MM. The investigators hypothesize that at a low tumor-burden disease, a lower dose of selinexor may be efficacious and lead to an improved toxicity profile than standard dosing.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Histologically confirmed diagnosis of SMM according to the IMWG definition: serum M-protein >/= 3 g/dL or BMPC >10% but <60%, or both.
* Should not meet CRAB criteria: hypercalcemia, anemia, bone lesions, or renal insufficiency thought to be related to the plasma cell disorder.
* Should have 1 of the following risk factors to be considered intermediate risk and 2 or more risk factors to be considered high-risk:
* BMPC>/=20%
* M-spike >/= 2g/dL
* Involved to uninvolved sFLC ratio of >/= 20
* normal hepatic function within 28 days prior to C1D1
* Adequate renal function within 28 days prior to C1D1. Estimated creatinine clearance (CrCl) calculated using formula of Cockcroft and Gault. CrCl >/= 15 mL/min.
* Adequate hematopoietic function within 28 days prior to C1D1: absolute neutrophil count (ANC)>/=1.5 x10^9/L, hemoglobin >/=10g/dL, platelets >/150x10^9/L.
* Life expectancy of >12 months.
* ECOG PS 0-1
* Subjects with reproductive potential must use 2 highly effective methods of effective contraception or practice sexual abstinence throughout the study and continue for 6 months after the study has closed. Subjects who are surgically sterile (e.g., history of bilateral tubal ligation, hysterectomy, or whos partner is sterile are not required to use additional modes of contraception.
* Ability to understand and willingness

Exclusion Criteria:

* Meets criteria for symptomatic MM as defined by any of the following, determined to be related to the plasma cell disorder

  * Hypercalcemia (corrected serum calcium >11.0 mg/dL)
  * Renal insufficiency (creatinine >2.0 mg/dL)
  * Anemia (hemoglobin <10g/dL)
  * One or more osteolytic bone lesions on radiography, but more than one lesion required if <10% clonal bone marrow plasma cells. Based on MRI imaging, there must be more than one lesion >5mm in size.
  * Clonal bone marrow plasma cells ≥60%
  * An involved serum free light chain ≥ 100mg/L with the ratio of the involved/uninvolved free light chains also ≥100
* Documented systemic light chain amyloidosis
* Systemic corticosteroids >10mg prednisone (or equivalent) daily for other medical conditions.
* Active invasive malignancy within the past 3 years that may affect the results or interfere with the interpretation of results of this study.
* Non-invasive malignancy that was not treated with curative intent within the past 3 years that may affect the results or interfere with the interpretation of the results of this study.
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within 14 days of the receiving the first dose
* Known active HIV infection without adequate anti-retroviral therapy
* Active gastrointestinal dysfunction that prevents patient from swallowing tablets or may interfere with absorption of study treatment
* Pregnant, breast feeding, or planning to become pregnant within 6 months after the end of treatment.
* Subject of reproductive potential that is not willing to use two methods of highly effective contraception during treatment period and for 6 months after the end of treatment.
* Any major medical or psychiatric disorder that, in the opinion of the investigator, might prevent the subject from completing the study or interfere with the interpretation of the study results.
* Prior exposure to a SINE compound, including Selinexor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of progression to Multiple Myeloma | 2 years after end of treament
  The study will assess how long participants will not have the cancer get worse while treated with selinexor

SECONDARY OUTCOMES:
Change in monoclonal protein (M-spike) or serum free light chains (sFLC) | 1 Year
  M-spike will be measured in g/dL and sFLC will be measured in mg/dL
Progression free survival | 1 Year
  The study will assess how long participants will not have the cancer get worse while treated with Selinexor
Rate of skeletal related events | 1 Year
rate of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Lipof, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No